CLINICAL TRIAL: NCT05866393
Title: Clean Hands Accessible and Manageable for Patients (CHAMPs): A Technology-based Self-management Intervention to Improve Patient Hand Hygiene and Reduce Hand Contamination Among Older Adults
Brief Title: Clean Hands Accessible and Manageable for Patients (CHAMPs)
Acronym: CHAMPs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Louis Stokes VA Medical Center (U.S. Federal Agency); MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Shanina Knighton, Research Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AG078273 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-05-19 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Pathogen Transmission; Patient Participation; Aging
Keywords: patient hand hygiene; self-management; infection prevention and control; older adult
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: In this 4-year project, the investigators will conduct a two-group parallel-design, RCT to determine the efficacy of a novel technology-based patient hand-hygiene system (CHAMPs) as a method to improve hand-hygiene behavior and reduce patients' hand contamination (Aim 1).
Masking Description: Using the randomization software the investigators will know who is in the CHAMPs or UC groups and will then assign the newly enrolled participant to an interventionist at each site. The randomization software will assign 0's and 1's. The 1's will indicate who is in the intervention group. For those assigned to CHAMPs, the interventionist after baseline data is collected will go in to set up the participants for the intervention which entails the CHAMPs system being placed on the bedrail and participants shown how it works and a patient return demonstration of use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Based on the literature reviewed and previous studies, the enrollment and the control group (Group 1- Usual Care) will begin within 24 hours of participants' admission to medical surgical units (4A, 4B, 5A, 5B- Cleveland VA and 9B, 9C, 11C, 7A MetroHealth). Data collection times are: the day of admission (Baseline, Day 0-1) and Day 3-4 between 2pm and 5pm. Participants will be consented for the research study staff to collect swabs for their nares on Day 0-1 and Day 3-4 and their hands at admission Day 0-1 and Day 3-4. No education or hand hygiene products will be provided. It is established that at both institutions a lemon towelette packet is provided with each meal.
- Clean Hands Accessible and Manageable for Patients (Experimental): CHAMPs participants will receive a patient hand-sanitation system attached via an R-shape clip to the bed rail. After it is placed on the bed rail, the personalized verbal electronic audio reminder with the RA's voice to insert the participants' name, " ____ it is (breakfast, lunch, dinner) time, please clean your hands." The times will be within an hour window of 7 a.m., noon, and 5 p.m. The CHAMPs system will be labeled "For Patient Use Only." The times were chosen around meal times because these times also are similar to around the time when medications are being administered. The hands can be a vector for germs to the face and mouth as shown in the literature. On Day 3 or 4 whichever comes later without anticipated discharge, the Interventionist will provide the evaluation of intervention questionnaires, clean the system turn it in to the project manager to retrieve SD card which contains the month, day, time, and number of system usages.
  Interventions: Behavioral: Clean Hands Accessible and Manageable for Patients

INTERVENTIONS:
Behavioral: Clean Hands Accessible and Manageable for Patients — Use of a patient-smart hand sanitation dispenser that provides reminders that are non-beeping reminders.
  Arms: Clean Hands Accessible and Manageable for Patients

SUMMARY:
This study proposes the novel use of a bedrail-affixed technology-based patient hand hygiene system with verbal and visual reminders to improve hospitalized older adults' self-management of hand hygiene practice, which in return reduces harmful germs found on older adult's hands that lead to infections.

DETAILED DESCRIPTION:
The investigators long-term goal to establish sustainable, patient-centered interventions at the patient level to engage patients in safety and prevention by offsetting barriers such as physical and sensory limitations that prohibit older adults from actively cleaning their hands independently. Unfortunately, older adults are at highest risk for infections and yet while hand hygiene is the single most important way to prevent the spread of infection, mechanisms for older adults to minimize personal risk for infections is often overlooked. Many contamination elements exist in hospital settings and for older adults encountering high-touch surfaces and medical devices that harbor pathogens that lead to infections will occur. However, without assistance, hand-hygiene practice rates are poor among hospitalized older adults' due to frailty, limited dexterity and mobility, cognitive limitations, and risk of falling, which prohibits independent use of visible hand- hygiene products (e.g., wall dispensers, towelettes, in-room sinks). New solutions are necessary. Therefore, in this proposal, the investigators have updated this investigator-developed, technology-enhanced patient hand hygiene system. Clean Hands Accessible and Manageable for Patients (CHAMPs), the investigator-developed and pilot tested bed rail-affixed hand-sanitizing dispenser, which features verbal, auditory and visual reminders to remind patients to sanitize hands. The safe and easily accessible motion-sensing system with usage tracking requires very little physical effort, as users need only to be able to freely move upper extremities and reach over to the bed rail to clean hands when prompted (e.g. before meal times). Pilot results among both a small group of older adults and in a high-tech simulated environment demonstrated both efficacy and feasibility of the intervention. In this 4-year project, the investigators propose a large heterogeneous randomized controlled trial (RCT) comparing two groups of hospitalized adults ≥ 65 years in two public hospitals, one group receives CHAMPs (n=125) and the other is the usual-care (UC) group (n=125). Study investigators consists of early and late stage investigators who have a successful record of working together and are ready to address the following aims: (1) to determine the effect of CHAMPs as a method to improve hand hygiene behavior and reduce patients' hand contamination, (2) assess the implementation of the intervention and (3) examine factors that influence outcomes associated with the intervention. The primary outcome is hand contamination as measured by presence, type, and quantity of colony forming units located on participants' hands. The research study staff's preliminary results offer promise that the CHAMPs technology-enhanced intervention may be an effective approach to engage patients in infection prevention as a solution to reduce colonization and infection rates among older adults.This proposal aligns with all four goals of NIH/NIA's 2020-2025 strategic plan, which is to improve the health, well-being, and independence of adults as age increases and to prevent or reduce the burden of age-related diseases, disorders, and disabilities.

ELIGIBILITY:
Inclusion Criteria:

1. > 65 years of age,
2. Admitted to a medical-surgical unit,
3. Expected to be hospitalized for more than 24 hours,
4. Written informed consent within 24-48 hours of admission, and
5. Speak and read English
6. Physical capacity to use the CHAMPs system
7. Sufficient hearing and seeing capacity to indicate understanding and use of the intervention.

Exclusion Criteria

1. terminal illness that prohibit interaction with CHAMPs
2. behavior disorder
3. violent behavior
4. physical or cognitive impairments that prohibit interaction with CHAMPs
5. limiting understanding and use of CHAMPs
6. undergoing radiation or chemotherapy that prohibit interaction with CHAMPs
7. skin disorders or
8. broken skin on hands.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient Hand Contamination Presence/Absence with Select Pathogens at Baseline | Day 0
  The primary effect of interest is that of the CHAMPs intervention on hand contamination at day 3-4 of study stay. The research study staff will test the presence/absence of hand contamination using a test of proportions that compares the two study arms using a two-sided test with an α = 0.05. > 1 colony forming unit of the following organisms susceptible to hand sanitizer: Enterobacteriaceae, Enterococci, Staphylococcus aureus, and Yeastis indicative of presence whereas 0 is indicative of absence. Colony forming units, or CFUs, are a unit of measurement used to determine the number of bacterial cells in a probiotic supplement or lab sample. CFU/ml is equal to the total number of colonies multiplied by the dilution factor and this is divided by the volume of the culture plate. CFU/ml - (Number of colonies*dilution factor) / volume of culture plate.
Patient Hand Contamination Presence/Absence with Select Pathogens at Day 3-4 | Day 3 or 4
  The primary effect of interest is that of the CHAMPs intervention on hand contamination at day 3-4 of study stay. The research study staff will test the presence/absence of hand contamination using a test of proportions that compares the two study arms using a two-sided test with an α = 0.05. > 1 colony forming unit of the following organisms susceptible to hand sanitizer: Enterobacteriaceae, Enterococci, Staphylococcus aureus, and Yeastis indicative of presence whereas 0 is indicative of absence. Colony forming units, or CFUs, are a unit of measurement used to determine the number of bacterial cells in a probiotic supplement or lab sample. CFU/ml is equal to the total number of colonies multiplied by the dilution factor and this is divided by the volume of the culture plate. CFU/ml - (Number of colonies*dilution factor) / volume of culture plate.
Patient Hand Contamination Counts of Pathogens at Baseline | Day 0
  The secondary effect retrieved after accomplishing presence or absence is the number of colony forming units (CFU) counts of pathogens. Participants with superior hand hygiene should have less multidrug-resistant organisms on their hands as measured by colony forming units when comparing baseline to the day 3-4 collection of hand swabs. Colony forming units, or CFUs, are a unit of measurement used to determine the number of bacterial cells in a probiotic supplement or lab sample. CFU/ml is equal to the total number of colonies multiplied by the dilution factor and this is divided by the volume of the culture plate. CFU/ml - (Number of colonies*dilution factor) / volume of culture plate.
Patient Hand Contamination Counts of Pathogens at Day 3-4 | Day 3 or 4
  The secondary effect retrieved after accomplishing presence or absence is the number of colony forming units (CFU) counts of pathogens. Participants with superior hand hygiene should have less multidrug-resistant organisms on their hands as measured by colony forming units when comparing baseline to the day 3-4 collection of hand swabs. Colony forming units, or CFUs, are a unit of measurement used to determine the number of bacterial cells in a probiotic supplement or lab sample. CFU/ml is equal to the total number of colonies multiplied by the dilution factor and this is divided by the volume of the culture plate. CFU/ml - (Number of colonies*dilution factor) / volume of culture plate.

SECONDARY OUTCOMES:
Patient Hand Hygiene Practice at Baseline | Day 0
  Secondary measure of hand hygiene practice will be indicated by hand sanitizer volume used. The bottle of hand sanitizer will be weighed before and after in milligrams (mg). Substracting the end weight from the baseline weight (mg) provides the weight which will then be converted into the difference in volume used. The equivalent of 1 Milligrams (mg) measurement of weight is equivalent to 1 Milliliters (ml) measurement of volume of liquid. The final measurement will be reported in milliliters (ml). Higher use of hand sanitizer volume indicates increased practice.
Patient Hand Hygiene Practice at Day 3-4 | Day 3 or 4
  Secondary measure of hand hygiene practice will be indicated by hand sanitizer volume used. The bottle of hand sanitizer will be weighed before and after in milligrams (mg). Substracting the end weight from the baseline weight (mg) provides the weight which will then be converted into the difference in volume used. The equivalent of 1 Milligrams (mg) measurement of weight is equivalent to 1 Milliliters (ml) measurement of volume of liquid. The final measurement will be reported in milliliters (ml). Higher use of hand sanitizer volume indicates increased practice.

CONTACTS AND LOCATIONS:
Overall Officials: Shanina C Knighton, PhD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - Lous Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No